CLINICAL TRIAL: NCT06407024
Title: Laparoscopic Versus Robotic Lateral Transabdominal Adrenalectomy: a Single-center Randomized Prospective Trial
Brief Title: Laparoscopic Versus Robotic Lateral Transabdominal Adrenalectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-422
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Adrenalectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 27 patients assigned to laparoscopic transabdominal adrenalectomy (Active Comparator)
  Interventions: Procedure: laparoscopic transabdominal adrenalectomy
- 27 patients assigned to robotic transabdominal adrenalectomy (Active Comparator)
  Interventions: Procedure: robotic transabdominal adrenalectomy

INTERVENTIONS:
Procedure: laparoscopic transabdominal adrenalectomy — Adrenalectomy performed by laparoscopic approach
  Arms: 27 patients assigned to laparoscopic transabdominal adrenalectomy
Procedure: robotic transabdominal adrenalectomy — Adrenalectomy performed by robotic approach
  Arms: 27 patients assigned to robotic transabdominal adrenalectomy

SUMMARY:
This study is being done to compare Laparoscopic vs Robotic lateral transabdominal adrenalectomy, these procedures are both standard of care.

The study team would like to compare both patient outcomes and surgeon efficiency and perspectives among both procedures.

The information from this study will help improve patient care, patient outcomes and maximize the appropriate utilization of resources in adrenal surgery.

DETAILED DESCRIPTION:
Adrenalectomy used to be done through big open chevron, subcostal or thoraco-abdominal incisions that led to significant recovery and morbidity. In 1990s, the description of laparoscopic adrenalectomy revolutionized the care of these patients by converting the procedure into a minimally invasive operation with a short hospital stay and recovery. Since then, many centers have reported the safety and efficacy of laparoscopic adrenalectomy. Laparoscopic surgery uses rigid, straight instruments operated by the surgeons under the visual guidance of a two-dimensional video platform.

In the late 2000s, robotic systems have been developed that incorporated articulating wristed instruments used with a three-dimensional computerized video platform. Over the past two decades, robotic systems have penetrated many thoracic, cardiac and abdominal procedures.

A review of the National inpatient database in 2016 showed that 32.7% of the adrenalectomies in the US are being done robotically and 48.5% laparoscopically. Nevertheless, there are scant comparative data and only two randomized studies comparing laparoscopic with robotic adrenalectomy, one of which suffers from a small sample size (10 patients in each group Morino et al Surg Endosci) and the other from exclusion of tumor types (pheochromocytoma only Ma W et al Eur J Surg Oncol). The first study found laparoscopic approach to be superior and the latter study robotic approach to be more advantageous. Both studies highlighted the cost of robotic surgery to be a disadvantage versus laparoscopic approach. Underscoring the lack of data to recommend one technique versus the other, a meta-analysis concluded that robotic adrenalectomy is a safe and feasible procedure with similar clinical outcomes as the laparoscopic approach and recommended high quality randomized clinical trials to determine whether laparoscopic vs robotic approach was superior to perform adrenalectomy.

The study team's clinic has a high-volume minimally invasive adrenalectomy program with a good mixture of laparoscopic and robotic surgical expertise, performing close to 100 surgical cases a year. There are a number of barriers to performing the randomized studies required for adrenalectomy. The first one is the adrenal surgery volume. An average general surgeon does one adrenal surgery a year. A high-volume adrenal surgeon is considered to do > 4-6 adrenalectomies a year. Furthermore, there are only a few centers in the world that possesses a large both laparoscopic and robotic adrenalectomy experience. Being a unique adrenal surgery center, the study team believes that their center is one of the few centers in the world qualified to perform a randomized clinical trial comparing laparoscopic with robotic adrenalectomy. The study team believes that such a study will help understand whether one approach is more advantageous over the other regarding surgical outcomes, especially with the increasing use of robotics in surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between ages 18 and 75
2. Diagnosis of an adrenal tumor/pathology planned for a minimally invasive adrenalectomy at the department of endocrine surgery at the Cleveland Clinic.

Exclusion Criteria:

1. Requirement for an open adrenalectomy based on imaging studies suggesting an aggressive cancer.
2. The presence of extensive surgical history precluding a minimally invasive approach to be undertaken.
3. Patients planned for a partial, rather than a complete adrenalectomy, as the former is a much easier procedure.
4. Patients planned for a posterior adrenalectomy (these would be patients with an extensive surgical history with significant intra-abdominal adhesions and those requiring bilateral adrenalectomy).
5. Mental incapacity or language barrier
6. Any condition, unwillingness, or inability, not covered by any of the other exclusion criteria, which, in the study clinician's opinion, might jeopardize the subject's safety or compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin-to-skin operative time | 1 day
  The duration of the procedure measured in hours and/or minutes

SECONDARY OUTCOMES:
Conversion to robotic or laparoscopic approach | 1 day
  The number of patients who are required to convert to either a robotic or laparoscopic approach - a departure from what they were randomized to.
Postoperative pain scores (according to visual assessment score 0-10, with 0 being non pain and 10 being worst pain) | 1 day
  Post operative patient pain ratings on a scale of 0 - 10
Hospital stay | 3 days
  Length of hospital stay as measured in days
Cost | 1 day
  Reported as disposable/reusable median cost ratio and operating room time-cost ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Eren Berber, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed internally and a manuscript will be prepared. Data is not planned to be shared with outside or other investigators